CLINICAL TRIAL: NCT05674032
Title: Detection of Causative Agents of Acute Pyelonephritis Using Bacterial Metallophores
Brief Title: Bacterial Metallophores in the Diagnosis of Acute Pyelonephritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Thomayer University Hospital (Other)
Collaborators: Czech Academy of Sciences (Other)
Responsible Party: Principal Investigator, Jan Hrbacek, M.D., Principal Investigator, Thomayer University Hospital
Other Study IDs: TUH00064190
Record Dates: First submitted 2022-09-22; First posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Acute Pyelonephritis; Complicated Urinary Tract Infection
Keywords: metallophores; mass spectrometry; acute pyelonephritis; complicated urinary tract infection; siderophores; yersiniabactin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cases: In-patients with AP or cUTI admitted for treatment to the hospital.
- Control group 1: Out-patients seeking treatment for uncomplicated acute cystitis.
- Control group 2: In-patients admitted to the ward without signs and symptoms of a urinary tract infection and with a negative urine culture result.

SUMMARY:
The project aims to investigate bacterial metallophores as potential diagnostic markers of acute pyelonephritis and complicated urinary tract infections. These secondary metabolites are excreted by pathogenic microorganims in the course of infection for the uptake of iron and other metallic ions from the host. They are species-specific and can be detected in body fluids (including urine) by mass spectrometry. The potential contribution of this project is a culture-independent method for the diagnosis of the causative microbiological agent.

DETAILED DESCRIPTION:
Acute pyelonephritis (AP) is a clinical syndrome characterized by fever, chills, nausea vomiting and costovertebral angle tenderness, bacteriuria and pyuria. The underlying pathophysiology is based on the presence of microbes in the renal parenchyma which may progress to sepsis. Complicated urinary tract infection (cUTI) is one accompanied by abnormalities of the urinary tract or host factors which make the eradication of the infection difficult.

The most common etiological agents include gram-negative enteric rods, i.e. E. coli, Klebsiella pneumoniae; and Enterococcus spp. Empirical antibiotic treatment should be targeted once culture and sensitivity results become available. This usually takes 24-48 hours, occasionally even 72 hours. Inadequate antibiotic treatment leads to higher mortality if the etiological agent is of a multi-drug resistant phenotype.

Metallophores are a major virulence factor of bacterial pathogens. These are chelating molecules secreted by the microbe for the uptake of iron, copper, and other metals from the host. E.g., siderophores aim at Fe3+ ions removal from the host protein molecules; the complex then adheres to specific extracellular receptors on the microbial cell and is internalized. Yersiniabactin is another metallophore which binds copper.

Proteomic analysis using mass spectrometry has been used in the detection of biomarkers for several pathological conditions: renal failure, post-transplant nephropathy, various malignancies etc. Metallophores can be detected by mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* in-patient with clinical signs and symptoms of AP/cUTI or out-patient with clinical signs and symptoms of acute uncomplicated pyelonephritis or in-patient with no clinical signs of UTI and a negative standard urine culture result

Exclusion Criteria:

* inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the department of urology and fulfilling eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-06-24 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Detection of metallophores | through study completion, an average of 1 year
  The detection of metallophores in urine samples
Classification of microorganisms | through study completion, an average of 1 year
  Taxonomic classification of the pathogenic microorganism using its metallophores

SECONDARY OUTCOMES:
Metallophores versus culture | through study completion, an average of 1 year
  The comparison of standard urinary culture results with those obtained from mass spectrometry analysis
Cases versus Controls 1 versus Controls 2 | 1 year after study completion
  The comparison of the detection of metalophores in cases with AP/cUTI versus acute uncomplicated cystitis versus urinary tract infection-free individuals

CONTACTS AND LOCATIONS:
Overall Officials: Jan Hrbacek, PhD., Study Director — Thomayer University Hospital
Locations (1):
- Thomayer University Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bonkat G, Bartoletti R, Bruyère F, Cai T, Geerlings SE, Köves B, et al. Guidelines on Urological Infections. 2020. Vallejo-Torres L, Pujol M, Shaw E, Wiegand I, Vigo JM, Stoddart M, et al. Cost of hospitalised patients due to complicated urinary tract infections: A retrospective observational study in countries with high prevalence of multidrug-resistant Gram-negative bacteria: The COMBACTE-MAGNET, RESCUING study. BMJ Open 2018;8:1-9. https://doi.org/10.1136/bmjopen-2017-020251. Hrbacek J, Cermak P, Zachoval R. Current antibiotic resistance trends of uropathogens in central europe: Survey from a tertiary hospital urology department 2011-2019. Antibiotics 2020;9:1-11. https://doi.org/10.3390/antibiotics9090630. Hyun M, Noh CI, Ryu SY, Kim HA. Changing trends in clinical characteristics and antibiotic susceptibility of Klebsiella pneumoniae bacteremia. Korean J Intern Med 2018;33:595-603. Caza M, Kronstad J. Shared and distinct mechanisms of iron acquisition by bacterial and fungal pathogens of humans. Front Cell Infect Microbiol 2013;4:1-23. https://doi.org/10.3389/fcimb.2013.00080. Prichystal J, Schug K, Lemr K, Novak J, Havlicek V. Structural analysis of natural products. Anal Chem 2016;88:10338-46. Václavková J, Ozdian T, Hajdúch M, Džubák P. Body fluids as a source of prote-omic biomarkers of various diseases. Chem List 2020;114:209-15 Skriba A, Pluhacek T, Palyzova A, Novy Z, Lemr K, Hajduch M, et al. Early and non-invasive diagnosis of aspergillosis revealed by infection kinetics monitored in a rat model. Front Microbiol 2018;9:1-7. https://doi.org/10.3389/fmicb.2018.02356. Hrbacek J, Morais D, Cermak P, Hanacek V, Zachoval R. Alpha-diversity and microbial community structure of the male urinary microbiota depend on urine sampling method. Sci Rep 2021;11. https://doi.org/10.1038/s41598-021-03292-x.